# Partners Human Research Committee Detailed Protocol

**TITLE:** Understanding and Improving Health Insurance Coverage among Long-Term Follow-Up Study Cohort Participants

PI: Elyse R. Park, PhD, MPH

**GRANT NUMBER:** RSGI-18-135-01 - CPHPS

VERSION DATE: 5/20/22

I. BACKGROUND AND SIGNIFICANCE

## a. Historical Background

Childhood Survivors are a growing population in need of medical surveillance. Children diagnosed with cancer have experienced improved survival rates over time, with more than three-fourths becoming long-term survivors. However, survivors of childhood cancer often face new and continued health care challenges and require ongoing care to monitor and treat long-term effects of their cancer and treatment throughout adulthood. Ongoing medical treatment and surveillance, with access to quality healthcare and coverage, are critical.

Although quality health insurance coverage is critical to this population, it has been complex to obtain. Given their ongoing health care needs, obtaining and navigating health insurance coverage is vital to ensure access to needed survivorship care. However, this can be difficult for individuals with pre-existing conditions such as a cancer diagnosis, who have historically faced denials of coverage, steep premiums, or "job lock" that keeps them from changing jobs for fear of losing coverage. 2,3 At the same time, childhood survivors have had higher rates of uninsurance, unmet health care needs, and burdensome costs. 4-10 These survivors are also less likely than siblings to be employed, married, and have a higher household income. 11-13 Dr. Park found that childhood survivors and siblings had similar rates of coverage, yet they differed by types of coverage and experiences obtaining coverage. 4 Uninsured survivors in particular were more likely to experience financial burdens from medical care that affected their care utilization.

Health care reform offers opportunities for childhood survivors to obtain quality coverage. The ACA<sup>14</sup> was signed into law in 2010 and is intended to increase access to affordable, quality health care. ACA policies offer considerable opportunities for populations with pre-existing conditions like childhood survivors to obtain coverage and improve access to needed care. Dr. Park and colleagues delineated the implications of specific ACA provisions for insurance coverage for childhood survivors.<sup>15</sup>

Although the ACA has increased coverage rates, uninsurance and underinsurance may remain a problem for childhood survivors. The ACA and other unprecedented changes to the health care landscape offer both opportunities and risk to childhood survivors regarding insurance adequacy and underinsurance. From Dr. Park's 2011-2012 CCSS (Childhood Cancer Survivor Study) health insurance survey we found that childhood survivors lacked awareness about the ACA<sup>16</sup> and had concerns that the ACA would increase their costs and threaten their quality and continuity of coverage.<sup>5, 16,17</sup> While the ACA requires coverage with no out-of-pocket costs for preventive services with "A" or "B" U.S. Preventive Services Task Force (USPSTF) ratings, these guidelines are not based on survivor-specific preventive guidelines and, as such, may not cover personalized screening recommendations.<sup>18</sup>

Limitations in health insurance literacy can make choosing and using health insurance challenging. With the complex and confusing array of evolving insurance designs, being able to understand and navigate insurance benefits is crucial for survivors to obtain the health care they need. However, many people have inadequate understanding of available insurance benefits and resources, and have limited health insurance literacy (i.e. perceived knowledge, ability, and confidence to make informed decisions about choosing and using health insurance). Vulnerable populations, such as those with low income and poorer health, are more likely to have limited health insurance literacy. Understanding specific insurance benefits and larger ACA policies may help survivors maximize coverage and prevent unmet need and burdensome costs.

Patient navigation interventions help patients overcome health care barriers. Patient navigation is a patient advocacy approach that was introduced in 1990, by Dr. Harold Freeman, to decrease high rates of breast cancer death among Black women in Harlem.<sup>28</sup> Patient navigation aims to reduce cancer disparities and negative health outcomes among vulnerable patient populations. Patient navigators were envisioned as proactive patient advocates who provided logistic and emotional support to promote patients' access to timely care.

**Existing navigator programs offer limited assistance with understanding and managing health insurance benefits and costs.** The US healthcare system is complex. Even with reform under the ACA, understanding insurance options remains complicated and a source of frustration for consumers. While addressing insurance barriers to accessing care may be a component of some navigator programs, navigators focused specifically on helping patients understand and use their insurance benefits are rare. Navigator services mandated by the ACA in health insurance exchanges are available to help consumers choose and enroll in coverage, but their reach does not extend beyond enrollment. Many exchange enrollees have sought navigation services post-enrollment to help understand their new insurance plans, but such post-enrollment services are unavailable. At the same time, cost-sharing under the ACA will continue to increase as coverage was not stabilized by Congress via payments to insurers to

reduce costs for consumers. Survivors in particular are going to need comprehensive assistance with insurance in future years.

#### b. Previous Studies

Childhood survivors and health insurance. In 2005 Dr. Park published findings in the Journal of Clinical Oncology demonstrating that CCSS survivors, compared to siblings, were significantly more likely to be uninsured and have difficulties obtaining health insurance.4 In 2009-2010 she conducted in-depth interviews with a subset of CCSS survivors<sup>2,5</sup> and with Drs. Kirchhoff, Donelan, and Kuhlthau found that survivors had low coverage expectations, had difficulties understanding how to utilize their coverage, and inevitably worried about future health care costs. This team surveyed a randomly selected sample of CCSS participants and siblings about their health insurance coverage and perspectives about the ACA.26,27 Survivors were significantly less likely to have employer-sponsored coverage (79.4% vs. 86.0%; p=0.04) and more likely to be covered by Medicaid/State (12.3% vs. 4.4%; p=0.002). 15.4% of survivors vs. 1.6% of siblings had recently been denied insurance (p<0.001). Survivors were more likely to borrow money to pay medical expenses (17.3% vs. 9.0% siblings; p=0.002) and not fill a prescription due to cost (15.7% vs. 9.0% siblings; p=0.02). Only 27.3% of survivors and 26.2% of siblings reported familiarity with the ACA. Concerns about the ACA included costs, decreased access to quality coverage, and employment. The majority of survivors, across different types of insurances, indicated strong interest in an insurance education program.

Recent study team reports of childhood survivors' underinsurance and its effects on financial burden and health care utilization. Dr. Kuhlthau led analyses describing patterns of health insurance coverage and care accessibility and affordability in an NHIS sample of adult childhood cancer survivors compared to adults without cancer during 2010-2014. Significantly more childhood survivors reported being uninsured, delaying medical care (24.7% vs 13.0%), needing but not getting medical care (20.0% vs 10.0%), and having trouble paying medical bills (40.3% vs 19.7%), compared to controls (ps<0.0001).<sup>28</sup> In 2017, Dr. Park and the study team published findings in JAMA Internal Medicine and JCO documenting that, compared to siblings, childhood survivors were significantly more likely to endorse indications of being underinsured, including being 84% more likely to borrow money because of medical expenses, 80% more likely to worry about being unable to pay for a needed treatment, and 74% more likely to worry they wouldn't be able to afford to fill a prescription. In addition, childhood survivors were more likely to report spending a higher percentage of their income on out-of-pocket medical costs. Survivors reported spending almost more than \$1000 annual out-ofpocket costs compared to siblings. A higher percentage of income spent on out-ofpocket medical costs was significantly associated with survivors' problems paying medical bills (OR, 8.9; 95% CI, 4.4 to 18.0); deferring care for a medical problem (OR, 3.0; 95% CI, 1.6 to 5.9); skipping a test, treatment, or follow-up (OR, 2.1; 95% CI, 1.1 to 4.0); and thoughts of filing for bankruptcy (OR, 6.6; 95% CI, 3.0 to 14.3).<sup>29,30</sup>

*Intervention and program development with childhood cancer survivors.* Dr. Park has studied the health behaviors and perceptions of childhood cancer survivors. <sup>31-34</sup>

She directed an NCI-funded trial to decrease smoking rates among 796 CCSS smokers that was found to be efficacious. The published a qualitative paper that had shaped the intervention, as well as a process evaluation paper which examined intervention characteristics associated with cessation success. Dr. Park also has extensive experience conducting qualitative research to inform survivorship program development. Dr. Kirchhoff is leading the development and testing of a childhood cancer survivor transition program with a focus on the provision of survivorship care plans for patients and families.

Health insurance and individuals with chronic conditions. Dr. Kuhlthau has extensive experience studying health insurance issues for individuals with chronic conditions, including Medicaid populations and groups with high expenditures. 40-51 She has also studied unmet need, a commonly used measure of underinsurance. 52-54 She conducted work on the private health insurance and work-life benefit systems for children with chronic conditions 55,56 which resulted in guides for employers, families, and state employees. Dr. Galbraith's work has demonstrated that children and families with chronic conditions are vulnerable to health insurance designs with high levels of cost-sharing and may reduce use of needed care due to cost. 57-59 Dr. Kirchhoff published on coverage gaps, financial burden, and medical costs, and their impact on access to care among childhood, adolescent and young adult cancer patients and survivors. 60-62

Effects of new insurance designs and health reform policies. Dr. Galbraith led one of the first studies of health insurance exchange plans, which documented problems for exchange enrollees with financial burden and unexpected costs; 63 this study also identified challenges with understanding and choosing plans for families, many of whom wished for greater assistance navigating plan options. 23 Dr. Galbraith has conducted studies of unmet health care need and financial burden among children and families with chronic conditions in high-deductible and other insurance plans. 59, 64-66 She has examined the impact of increased cost-sharing on health care decision making and use of recommended health care services. 67-72 She is conducting a trial to evaluate how a price transparency tool can help high-deductible plan enrollees manage costs.

**Peer counselor and navigator-based interventions.** Dr. Park directed a smoking cessation trial, in collaboration with the Long-Term Follow-Up (LTFU) study at St. Jude Children's Research Hospital, in which she trained childhood cancer survivors to be smoking cessation peer counselors and deliver a phone-based intervention. <sup>32</sup> Dr. Galbraith conducted a randomized trial of a patient navigator intervention to reduce readmissions for high-risk patients discharged from a safety-net hospital. <sup>72,73</sup> Dr. Donelan has conducted extensive survey research examining patient barriers to cancer screening and follow-up and physician referral communication with patients. <sup>74-77</sup> She examined the effectiveness of a patient navigation program in improving minority patients' follow-up of an abnormal mammogram.

#### c. Rationale of Proposed Research

Health care reform under the Patient Protection and Affordable Care Act (ACA) offers considerable opportunities for childhood cancer survivors to obtain coverage and improve access to needed care. However, in the general population, many people have low understanding of available insurance benefits and resources, and have limited health insurance literacy (i.e. perceived knowledge, ability, and confidence to make informed decisions about choosing and using health insurance). Misperceptions about which services require out-of-pocket costs may lead some enrollees to avoid services that are in fact exempt from cost sharing. Even with coverage protections from the ACA, barriers to obtaining quality coverage (e.g., in states without Medicaid expansion) and accessing needed care may remain for childhood survivors. Understanding and navigating insurance benefits is crucial for cancer survivors to obtain the health care they need. In this new post-reform landscape, the degree to which coverage and costs have changed for childhood cancer survivors is still largely unknown.

## d. Study Site Roles

The sites in this study, MGH, St. Jude Children's Research Hospital, and the University of Utah will each have different, complementary roles. The Partners IRB will be the IRB of record for this study, and the collaborating IRBs of St. Jude and the University of Utah will CEDE review to the Partners IRB. Site and IRB roles are described below.

#### **MGH Site Roles**

As the IRB of record and lead site for this study, MGH will be responsible for the development and regulation of all study-related materials, documents, assessments, and interventions. For Phase 1 of the study, MGH will be specifically responsible for the facilitation of advisory board and participant focus group interviews, and the qualitative analysis this data. Utilizing the data garnered from these interviews, MGH will further develop and tailor the intervention content (though MGH will work with collaborators on this aspect of the study, MGH will lead in the development and final submission of this piece).

For Phase 2 of the study, MGH will be responsible for the delivery of the intervention content. Through the platform of MGH telehealth (Zoom), approximately 40 intervention arm participants (recruitment processes are described below) will receive brief health insurance educational sessions by a health insurance navigator. MGH will be responsible for the training and supervision of the navigator.

For Phase 3 of the study, MGH will be responsible for the facilitation and analysis of exit interviews conducted with the Phase 2 intervention arm participants (MGH will not be conducting the exit interviews. See University of Utah Phase 3 roles for more information).

#### St. Jude Site Roles

As one of the collaborating sites for this study, St. Jude will be responsible for all recruitment activities. St. Jude Children's Research Hospital is the site of the Long-Term Follow-up Study (LTFU), and study participants will be exclusively recruited from the

eligible members of this cohort. St. Jude will be responsible for recruiting, randomly selecting, and consenting participants for the focus group interviews, the open pilot of the study intervention, and the pilot randomized trial. Once recruited and consented, St. Jude will securely send relevant participant information to the study staff at the University of Utah and MGH.

## **University of Utah Site Roles**

As one of the collaborating sites for this study, the University of Utah will be responsible for all participant assessments during the study. During Phase 1 of the study, after receipt of participant information from St. Jude, the University of Utah will coordinate with MGH to set up and schedule participant focus groups. For the open pilot of the study, St. Jude will distribute baseline and follow up surveys to participants and will lead all quantitative analyses of these assessments. Lastly, the University of Utah will schedule and facilitate exit interviews with all open pilot participants and will securely send qualitative data to MGH for analysis. The University of Utah will also be responsible for remuneration of subjects during all phases of the study.

For Phase 2 of the study, the University of Utah study roles mirror those of Phase 1, with the distribution of baseline and follow-up surveys to participants, and the collection and analysis of said data.

For Phase 3 of the study, the University of Utah and MGH will coordinate to schedule exit interviews with the Phase 2 intervention arm participants.

#### II. SPECIFIC AIMS

## <u>Aim 1:</u> To develop a psychoeducational health insurance navigation program (HINP).

<u>A1a:</u> To qualitatively assess LTFU participants' reports of 1) barriers to accessing and using quality health insurance2) resources to support health insurance access and use, 3) navigation program content, 4) intervention structure and dose, 5) program delivery, 6) program acceptability, 7) aspects of coverage that are not well understood <u>A1b:</u> Aim 1b: To qualitatively assess approximately 3 advisory boards' and approximately 10 individual experts' feedback 1) barriers, 2) resources, 3) content, 4) intervention structure and dose, 5) delivery and 6) selection criteria <u>A1c:</u> To pilot the intervention with LTFU participants (approximate n=10).

## <u>Aim 2:</u> To conduct a <u>videoconferencing-based</u> pilot randomized trial of the HINP (n= approximately 80).

<u>A2a:</u> To assess the <u>feasibility</u> (number of eligibles enrolled and sessions completed) and <u>acceptability</u> (satisfaction, perceived support) of participants undergoing the HINP.

<u>A2b:</u> At 3-month post-program follow-up, to assess the efficacy of the HINP to assist participants with accessing and utilizing coverage and managing costs. Primary

outcomes are 1) health insurance literacy and 2) financial distress related to medical costs

<u>A2b Hypothesis:</u> The HINP, compared to enhanced usual care, will improve participants' health insurance literacy and decrease financial distress.

## Aim 3: To refine the HINP program for future use.

<u>A3a:</u> To explore HINP intervention arm participants' 1) satisfaction with the intervention, 2) recommendations for modifications on delivery modality, and 3) recommendations for intervention topics and content modifications.

**Study Design Overview:** The proposed study will take place in 3 phases and will involve a total of approximately 122 participants recruited from the Long-Term Follow-Up (LTFU) study cohort (See Section III below)-

- In Phase 1 we will develop a psychoeducational health insurance navigation program (HINP) through participant input and a series of advisory board meetings and individual interviews. We will also refine the program by recruiting a small group of LTFU study cohort members for an open pilot of the intervention.
- In Phase 2 we will pilot the feasibility, acceptability, and preliminary efficacy of the videoconferencing-based HINP with LTFU study cohort members.
- In Phase 3 we will further refine the program through study participant feedback.

Below we describe the activities for the three study phases. Detail on participant enrollment and consent procedures for all three phases is included in Section IV.

#### Phase 1

#### Participant Focus Groups

Four focus group interviews (approximately n=8 per group) will be conducted with randomly selected LTFU study participants (see Participant Focus Group Interview Guide); selection will be stratified according to Medicaid expansion status (Y/N), which we will determine based on participant demographic information from the LTFU data records. LFTU participants from the original and expansion cohort will be eligible and consented (Please refer to Sections III and IV for information on subject selection and consent procedures); we will assure inclusion of men and women. Groups will last about 60 minutes, and may be conducted through Zoom, a HIPAA compliant videoconferencing platform (see Maintaining Confidentiality in Section VII) or in-person. Participants will be provided \$50 remuneration by the University of Utah. Groups will be co-facilitated by co-investigators via a semi-structured interview guide (See Participant Focus Group Guide). The interviews will be recorded.

#### Advisory Board Input on HINP

Three advisory board meetings will be conducted, specifically, with national oncology clinicians and researchers and Boston-based experts. These groups will be cofacilitated by investigators via a semi-structured interview guide that contains the following domains: 1) barriers, 2) resources, 3) content, 4) intervention structure and

dose, 5) delivery and 6) selection criteria (See Advisory Interview Board Guide). Advisory board meetings will also be conducted through Zoom Videoconferencing, via phone, or in person. The advisory board focus groups will be recorded and used for quality improvement purposes of the HINP.

## **Expert Individual Interviews**

We will conduct approximately 10 30-minute individual interviews with experts at the intersection of health insurance, navigation, cancer, and survivorship. Experts will include clinicians, oncology social workers, and health insurance specialists. Interviews will be recorded and used for tailoring and improvement of the HINP. Individual interviews will be facilitated by investigators using a semi-structured interview guide containing the same domains as the advisory board interviews. These interviews will also be conducted through Zoom Videoconferencing via phone, or in-person.

For both Advisory Board and Expert interviews, we will assent experts for participation in the interviews (See Advisory Board Interview Guide)

## Qualitative Analyses to Inform HINP Development

For qualitative analyses of focus group, advisory board meetings, and individual interviews, all data will be analyzed by MGH and Utah study staff using NVivo qualitative software. Content analyses will be conducted including a structural thematic framework, categories, and coding plan. For focus group data, a coding framework will be developed for themes and codes according to participants' feedback on 1) barriers to accessing and using health insurance 2) resources to support health insurance access and use, 3) navigation program content, 4) intervention structure and dose, 5) program delivery, 6) program acceptability, 7) aspects of coverage that are not well understood (See Participant Interview Guide) For advisory board and individual interview feedback, a coding framework will be developed for themes and codes according to the domains of: 1) barriers, 2) resources, 3) content, 4) intervention structure and dose, 5) delivery and 6) selection criteria. To ensure coding reliability, coding discrepancies for participant focus groups will be resolved through discussion and comparison of raw data. Coding will continue until a high level of reliability (Kappa= >0.80) is established. Co-investigators will provide an expert review of the results. For expert and advisory board interviews, a Rapid Analysis method will be used.

## Open Pilot with Participants

With feedback from the focus groups, advisory boards, and individual interviews, results will be interpreted, summarized, and finalized; the investigators will refine the HINP. Then, approximately 5-10 participants will be randomly selected to participate as pilot subjects (Please see Sections III and IV for information on subject selection and consenting procedures). Aspects of the study that will be piloted include the surveys, intervention, and exit interview. Participants will be remunerated \$20 for the completion of a baseline survey, a follow-up survey and the exit interview by the University of Utah. Final intervention and survey modifications will be made.

#### Phase 2

## Pilot Trial Design

We will recruit and randomize approximately 80 LTFU participants to a health insurance navigation intervention or to enhanced usual care (Please see Sections III and IV for information on subject selection and consenting procedures). We have selected this sample size of approximately 40 per arm to enable evaluation of feasibility and acceptability goals as well as explore meaningful differences in the outcomes. Surveys will be conducted at baseline and 3-month post program completion follow-up via REDCap or mail. All participants will be asked to complete a follow-up survey approximately 3-months after the HINP intervention period (in other words approximately 5-months post pilot trial enrollment).). After completion of the follow-up survey, HINP participants will be contacted for an exit interview (see Phase 3 below). Participants will be remunerated \$20 for each survey and the exit interview by the University of Utah

## Study Arms

#### Enhanced Usual Care

Enhanced usual care will consist of a mailed or online copy of a health insurance resource guide.

## Navigation Intervention

The intervention will be delivered via synchronous videoconferencing (real-time delivery and communication between the navigator and the participant) by a trained patient navigator (See Intervention Fidelity in Section VI) and will consist of 4, 30-minute sessions delivered every week, over the span of one month (for intervention development purposes, the pilot sessions will occur every week, over the course of one month). The navigation intervention group will also receive a mailed copy of the brochure.

## Proposed Navigation Intervention Structure and Content

The program will be delivered via videoconferencing by a navigator over a 1-month period. Accordingly, patient navigation is delivered until the desired endpoint is achieved; we propose that this will be accomplished with 4 navigation sessions (See Table 1: Proposed HINP Intervention). The proposed program content was informed by: 1) aforementioned research identifying childhood survivors' difficulties with accessing and utilizing one's coverage and managing costs, 2) CCSS health insurance survey, and 3) ACA provisions that are relevant to survivors (e.g., prevention services exempted from cost sharing, sources of available coverage and eligibility, benefits policies that have cost-related implications like OOP costs, and essential health benefits such as prescription medications. Based on advisory board and individual interview feedback, the content and tailoring of information will be modified.

## **Table 1: Proposed HINP Intervention**

**Session One: Learning About Survivorship Healthcare Needs** 

Sessions Two: Learning About Your Plan in Relation to Policy

Session Three: Navigating One's Own Plan

#### Phase 3

#### **Exit Interviews**

For HINP participants after the follow-up survey, the study co-investigators will conduct in-depth interviews (see Participant Exit Interview Guide) via videoconferencing with the 40 intervention participants to assess survivors' 1) satisfaction with the intervention, 2) recommendations for modifications on overall session topics and intervention content (e.g., physician communication, cost management strategies). and 3) recommendations for modifications on delivery modality (e.g., number and length of sessions, videoconferencing delivery). These will last about 20 minutes and participants will be remunerated \$20 for their time by the University of Utah. The exit interviews will be recorded.

Exit interview data will be transcribed and analyzed using NVivo qualitative software. Content analyses will be conducted and co-investigators will provide an expert review.

#### **III. SUBJECT SELECTION**

#### Participants: Inclusion and Exclusion Criteria

LTFU study staff at St. Judy Children's Research Hospital keep updated participant contact records for this study, which allows for participants to be approached for additional research studies. For Phases 1 and 2, the LTFU study staff will recruit a total of approximately 122 participants from the Long-Term Follow-Up Study cohort. Phase 1 will involve recruitment of 32 participants for four focus groups and approximately 5-10 participants for the open pilot. Phase 1 participants will not be eligible for Phase 2 participation. For the focus group activities of this Phase, participants will be randomly selected stratified according to whether they reside in a state with or without Medicaid expansion, which LFTU staff will determine based on participant addresses available from the LTFU data records.

Phase 2 will involve recruitment of 80 randomly-selected participants for the pilot randomized trial. Participants will be randomly selected stratified according to whether they reside in a state with or without Medicaid expansion, which LFTU staff will determine based on participant addresses available from the LTFU data records.

Phase 3 participants will be recruited from the Intervention Arm of Phase 2 (approximately n=40).

For both Phases, we will exclude participants who: (1) do not have health insurance, (2) are under the age of 18, (3) are unable to give informed consent due to psychiatric or cognitive impairment as determined in consultation with study PI, patient navigator, or oncology social worker, and (4) do not have access to an smartphone, computer or tablet with internet access. Importantly, we will closely document and monitor the

numbers of individuals who are unable to participate given this final criterion, as it will further inform the feasibility of this intervention modality.

## Sources of Subjects and Recruitment Methods

The Long-Term Follow-Up Study (LTFU) is an NIH-funded multi-institutional study of individuals who were diagnosed before 21 years of age with leukemia, CNS malignancies, Hodgkin's disease, non-Hodgkin's lymphoma, Wilm's tumor, neuroblastoma, soft tissue sarcoma, bone cancer or serious illness who survived at least five years after diagnosis. Eligible participants for the LTFU were identified through medical records and clinic lists at participating centers in the U.S., yielding a retrospectively ascertained cohort of adult childhood survivors with ongoing, longitudinal follow-up. The LTFU includes individuals diagnosed with cancer or serious illness between 1970-1999, recruited from over 25 pediatric oncology institutions in North America. Eligible participants for our study include 21,841 LTFU participants who are still alive and have available contact information.

#### IV. SUBJECT ENROLLMENT

#### Methods of Enrollment

Prospective participants for each phase of the study from the LTFU study cohort will be identified via LTFU records and recruited and consented at the CCSS Coordinating Center at St. Jude Children's Research Hospital (Supporting Facility for the LTFU) by LTFU staff. Prospective participants will receive an invitation to the study through email and mail (See LTFU Focus Group, Open Pilot, and Pilot Intervention Recruitment Letters). CCSS participants have consented to be contacted by the study and agreed to email communication by voluntarily providing us with their email address. St. Jude employs a system called Emma to administer and deliver email campaigns. Emma (myemma.com) is a secure email marketing platform that allows for multi-level campaigns with all or segments of our participants. It allows for contact management, simple HTML template design with piping and logical integration, tracking of email campaign receipts, errors, and opt-outs, and drilling down to review participant level activity If eligible and interested, prospective participants will read over an enclosed Research Consent Form, which they will have the option to either fill out via an online DatStat survey link (the system that St. Jude Children's Research Hospital uses for LTFU consenting procedures, see Data Management in V. Study Procedures) or to fill out the hard copy of the form and mail it back to LTFU staff at St. Jude Children's Research Hospital. Additionally, participants may also be recruited through telephone, with outreach being done by CCSS Coordinating Center, and a mailed version of the recruitment letter might be sent out, with instructions being provided for how to access the online consent portal. Potential participants will also be able to get more information about the study via a St. Jude website (which will also have a link to the online consent form). Following consent, the assignment of a unique study identification number to each participant, and randomization into intervention vs. control arms for Phase 2, participant information will be sent securely to Dr. Kirchhoff via SharePoint, an encrypted system used to transfer data. Dr. Kirchhoff's team will lead the focus group scheduling and survey facilitation, while both MGH and University of Utah study staff will coordinate the navigation intervention. The study interventionist may contact consented participants via telephone and email in to schedule intervention sessions.

#### Informed Consent

For the participant focus groups, open pilot, and pilot trial, informed consent will be facilitated by LTFU study staff using an IRB approved consent form for each piece of the study (See Focus Group, Open Pilot, and Pilot Intervention Consent Forms. The consent form will describe the study in detail, including the purpose of the research, clinical procedures, risks and discomforts, benefits, reimbursements, and alternatives to participation. Confidentiality, the right of each subject to request further information, and the right of each subject to withdraw from the study at any time, is fully detailed in each consent form. Patients will be informed via the consent form that they can freely choose not to participate. We will exclude participants who, as determined by the study PI or navigator, are unable to give consent due to psychiatric or cognitive impairment. There will be two separate consenting procedures for Phase 1 of the study. One consenting procedure will be for the focus group participants (n=32), and one consenting procedure will be for the open pilot participants (n=10). For Phase 2 of the study, there will be a single consent form for the pilot randomized trial participants (n=80). The intervention arm participants of Phase 2 (n=40) constitute the Phase 3 participants, so they will be consented for Phase 3 during the Phase 2 consent process. There will be separate consent forms that correspond to the described procedures.

## Intervention Assignment and Randomization

#### Pilot Trial

The CCSS Coordinating Center LTFU study staff will randomly select 80 participants among the LTFU cohort (original and expanded together). To do this, CCSS will use stratified random sampling, where we will divide the sample of LTFU participants into two groups: residing in a Medicaid expansion state or not. Random samples will then be selected from each of the two strata until 80 participants are consented and enrolled. The 80 selected participants will be randomized to either enhanced usual care (n=40), or the health insurance navigation intervention (n=40). After obtaining informed consent, participant information will be sent securely to Dr. Kirchhoff via SharePoint, an encrypted system used to transfer data. Dr. Kirchhoff's team will lead the pilot trial procedures.

## V. STUDY PROCEDURES

| | Recruitment and consent | Scheduling activity | Procedures | Data - qualitative | Data –<br>quantitative |
|---|---|---|---|---|---|
| Phase 1 | | | | | |
| Focus<br>groups | LTFU staff identifies Medicaid vs. not Medicaid from LTFU records; | Kirchhoff team receives consented list from LTFU via SharePoint; they set up FG time | MGH runs FG via<br>Zoom; records<br>and transcribes<br>the data | Per grant -<br>Content analyses<br>will be conducted<br>by Drs. Park and | None collected |

| | Randomly selects and consents Goal: 4 FG x 8 people -> 32 or so participants | working with MGH team to schedule | | the research assistant | |
|---|---|---|---|---|---|
| Open<br>pilot | LTFU staff randomly selects & consents participants Goal: 5-10 participants | Kirchhoff team<br>received<br>consented list<br>from LTFU via<br>SharePoint;<br>Kirchhoff team set<br>up sessions with<br>navigator | Kirchhoff team<br>collects baseline<br>and FU surveys<br>via REDCap | Dr. Park and or/<br>study navigator<br>and research<br>assistant will<br>conduct analyses | Per grant - Dr. Kirchhoff will lead the analyses of surveys; will receive additional data from LTFU study as needed (demographics, etc) via SharePoint |
| Phase 2 | - | | | | |
| Pilot | LTFU staff identifies Medicaid vs. not Medicaid from LTFU records; Randomly selects; Randomizes Participants after they consent Goal: 80 participants | Kirchhoff team receives consented list from LTFU via Sharepoint; Kirchhoff team set up sessions with navigator | Kirchhoff team<br>collects baseline<br>and FU surveys<br>via REDCap | None collected | Per grant - Dr. Kirchhoff will lead the analyses of surveys; will receive additional data from LTFU study as needed (demographics, etc) via Sharepoint |
| Phase 3 | | | | | |
| Exit<br>interviews | No new recruitment | Kirchhoff team will<br>help schedule the<br>interviews | Exit interviews run<br>by Utah team | Content analyses will be conducted by Drs. Park and Galbraith | None collected |

## Data Management, Collection, and Transfer

#### Recruitment

During the recruitment periods of each phase of the study, St. Jude will track and obtain consent through DatStat, which allows researchers to configure online mobile responsive web surveys with tailored logic checks and requirements, data prepopulating and piping, and portal access for quick reporting, analytics, and downloads. The system is HIPAA compliant and fully validated for 21 CFR Part 11. Once participants are consented to the study, their information will be sent to Dr. Kirchhoff and her team at the Huntsman Cancer Institute at the University of Utah via SharePoint. SharePoint is a secure file sharing service supported by the Huntsman Cancer Institute that is encrypted and HIPAA certified. It is password protected and Dr.

Kirchhoff's SharePoint file sharing can only be accessed by other investigators through invitation to ensure data privacy.

## **Quantitative Data**

For the pilot trial, Dr. Kirchhoff's staff at the Huntsman Cancer Institute at the University of Utah will oversee the scheduling participants and will ensure the completion of the baseline survey and follow-up surveys for both Phase 1 and 2 of the study. Survey data will be collected via a secure web-based portal (REDCap). REDCap is maintained by the bioinformatics shared resource at the Huntsman Cancer Institute where Dr. Kirchhoff is an investigator. As such, she has access to survey and database support for REDCap for all data collection activities. Data transmissions will occur between Dr. Kirchhoff and the CCSS Coordinating Center and Statistics and Data Center via SharePoint to facilitate data access from the LTFU baseline and follow up surveys for inclusion in the statistical analysis (https://ccss.stjude.org/documents/original-cohort-questionnaires). Dr. Kirchhoff will lead the pilot study survey data management and analyses, and transmit analytic data to MGH using SharePoint. Data will be managed and cleaned by Dr. Kirchhoff's data manager and overseen by Dr. Kirchhoff.

## Focus Group and Exit Interview Qualitative Data

Once the focus groups are scheduled by Dr. Kirchhoff's team, the data collection efforts will be led via MGH's Zoom program. The Phase 1 participant qualitative data will be collected and stored within MGH. Data will be collected by Dr. Park's team at Massachusetts General Hospital using recording devices. Audio recording files will be saved and uploaded into NVIVO software on Shared File Areas in the Partners network, which will only be accessible to IRB-approved study staff. NVIVO files will be sent securely via Partners Secure File Transfer or via SharePoint, which has been approved for use in this study. The Phase 3 qualitative data in the form of exit interviews will follow procedures detailed in Phase 1.

#### Advisory Board and Expert Interview Qualitative Data

After expert and advisory board interviews have taken place via Zoom, audio recordings will be stored on Shared File Areas in the Partners Network. Audio recordings will be directly uploaded into NVIVO and sent securely to study staff at the University of Utah for analysis.

## Intervention Arm Components

Of the approximately 80 participants recruited for Phase 2 of the study, 40 will be randomized to enhanced usual care, and 40 will be randomized to the health insurance navigation intervention. As described above, the intervention arm will involve 4 sessions delivered by a navigator.

#### Intervention Fidelity

The patient navigator (PN) will undergo training by the Co-investigators and pilot sessions. The NCI, with support from the ACS, established the Patient Navigation Research Program (PNRP) to implement and evaluate patient navigator programs. The PNRP developed a navigation performance checklist with 3 quality indicators of care:<sup>79,80</sup> 1) participant interaction (e.g., established rapport), 2) care management (assessed subjects' understanding), and 3) intervention delivery (e.g., relevant information provided on insurance options, cost savings). Study investigators will review 15% of patient navigation encounters using these quality indicator criteria.

#### Assessments

#### Phase 1 Assessments

During the Open Pilot of the intervention, participants will complete a baseline survey and a 3-month post-program follow up survey. Participants will be remunerated \$20 for the completion of each survey by the University of Utah. LTFU extracted medical record data will provide information on cancer diagnosis, age at diagnosis, years since diagnosis, and type of treatment. The open pilot will also involve an exit interview, which is described in further detail below.

## Phase 2 Assessments

During the pilot trial, participants will complete a baseline survey, a 3-month post-program follow up survey. LTFU extracted medical record data will provide information on cancer diagnosis, age at diagnosis, years since diagnosis, and type of treatment.

#### Phase 3 Assessments

After the completion of the follow-up survey, investigators will conduct In-depth exit interviews with the 40 intervention arm participants to assess participants' 1) satisfaction with the intervention, 2) recommendations for modifications on overall session topics and intervention content (e.g., physician communication, cost management strategies) and 3) recommendations for modifications on delivery modality (e.g., number and length of sessions, videoconferencing delivery). Participants will be remunerated \$20 for their time by the University of Utah.

#### VI. BIOSTATISTICAL ANALYSIS

#### Analysis Plan

## **Qualitative Data**

For qualitative analyses of participant focus groups advisory board meetings, individual expert interviews, and exit interviews, all data will be analyzed by MGH and University of Utah study staff using NVivo qualitative software. For qualitative analysis of advisory board and individual expert interviews, audio files will be uploaded into NVIVO software and analyzed using a Rapid Analysis method. Content analyses for the participant focus groups an exit interviews will be conducted including a structural thematic framework, categories, and coding plan. For focus group data, a coding framework will be developed. To ensure coding reliability, coding discrepancies will be resolved through

discussion and comparison of raw data. Coding will continue until a high level of reliability (Kappa= ≥0.80) is established. Co-investigators will provide an expert review of the results.

Focus Group Data: A coding framework will be developed for themes and codes according to participants' feedback 1) barriers to accessing and using health insurance 2) resources to support health insurance access and use, 3) navigation program content4) intervention structure and dose, 5) program delivery, 6) program acceptability, 7) aspects of coverage that are not well understood Advisory Board and Individual Interview Data: A coding framework will be developed for themes and codes according to the advisory board feedback on 1) barriers, 2) resources, 3) content, 4) intervention structure and dose, 5) delivery and 6) selection criteria

Exit Interview Data: A coding framework will be developed for themes and codes according to participants' feedback on 1) satisfaction with the intervention, 2) recommendations for modifications on overall session topics and intervention content (e.g., physician communication, cost management strategies). and 3) recommendations for modifications on delivery modality (e.g., number and length of sessions, videoconferencing delivery)

## Quantitative Data

For quantitative data, Dr. Kirchhoff's team at HCI will conduct the analyses with input from Dr. Park and her study team, and the LTFU study team. As discussed in Participants, we will sample by Medicaid expansion vs. non-expansion states. All analyses will be weighted using inverse sampling probabilities so that results are representative of the overall LTFU study cohort.

At baseline, all pilot participants will complete a baseline. The HINP navigator will use each participant's baseline survey responses to personalize and individualize sessions. At the 3-month post-program follow-up, participants will complete the Phase 1 survey Outcome questions, which will be asked within the 5-month time frame period after trial enrollment. Participants will also be asked questions below about feasibility and acceptability.

We will use descriptive statistics to report on the following endpoints: intervention feasibility (percent of participants enrolled), acceptability (satisfaction, perceived support) and efficacy (e.g., ACA familiarity, health insurance literacy, intention to adhere to recommended survivorship care, provider communication, and coverage status). Descriptive statistics will examine group differences at baseline; any imbalances will be adjusted. We will use chi square and independent t-tests to compare end-of-intervention changes in preliminary efficacy outcomes between the two groups. Although a 3-month post intervention follow-up period is brief, we will also conduct exploratory comparisons with other study outcomes to see if trends change in the expected direction. We will compare pre/end-of-treatment, within groups, with paired t-tests. In addition, we will use bivariate statistics to examine sociodemographic and cancer-related factors (type of

diagnosis, age at diagnosis, years since diagnosis, cancer treatment, chronic conditions<sup>81</sup>, cancer treatment (e.g., cranial radiation yes/no, anthracycline exposure yes/no) associated with feasibility, acceptability and preliminary efficacy outcomes.

## <u>Outcomes</u>

## Primary Outcomes: Feasibility and Acceptability.

1. Feasibility: Number of eligible enrollees and number of sessions completed. 2. Acceptability: 4-point scales of satisfaction with navigation services (To what extent has this program met your needs? Did you get the kind of health insurance assistance that you wanted? How helpful has this program been for you?) and perceived support (emotional/informational scale of the Medical Outcomes Study social support survey, an 8-item scale widely used with cancer patients). 82-86

## Secondary Outcomes: Efficacy.

The ACS's National Patient Navigator Leadership Summit recommend patientnavigation outcome measures, which included: perceived knowledge, perceived confidence in overcoming barriers to care, and satisfaction with patient navigation services. Accordingly, we will measure: 1) health insurance literacy, 2) financial distress related to medical costs.

3) familiarity with healthcare reform policies, 4) insurance status (among those insured at study enrollment), and 5) discussion with providers about health care costs<sup>63</sup> and preventive services among those having a visit during this interval (2-item y/n questions).

#### Measures

To evaluate the pilot, we will use a mixed methods data collection approach, using both quantitative survey items and open-ended questions. <sup>87</sup> Most study measures will come from survey questions repeated from the 2011-2012 CCSS health insurance survey (see Appendix); some new questions will be added and are indicated as such. Survey development included a qualitative study conducted with a sample of LTFU participants, <sup>5</sup> modifications and inclusions of national survey questions <sup>87-92</sup> and a cognitive testing phase. Using data collected previously by the overall LTFU via abstraction of medical records, data will be used to provide information on cancer diagnosis, age at diagnosis, and cancer treatment. These data will be provided to Dr. Kirchhoff's team via SharePoint, an encrypted system used to transfer data. Data from the LTFU surveys will provide information on sociodemographic and medical history since cancer treatment, and presence of a medical late effects and chronic health conditions including second cancers. The measures will include the following:

#### Participant Characteristic Measures (see study surveys)

Characteristics: Age, Gender, Education, Race/Ethnicity, Partnership/Marital Status

Enabling Characteristics: State of Residence, Familiarity with ACA Policies

Health Insurance Literacy: Confidence in Understanding of Terms (e.g. Coinsurance), Confidence in Choosing, Comparing, and Using Insurance, Household and Personal Income

Need: Cancer Diagnosis, Age at Diagnosis, Years Since Diagnosis, Treatment Type, Recurrence of Primary Cancer, Second Malignancy, Other Chronic Conditions.

#### Outcome Measures

Insurance Coverage: Insurance Status, Difficulty or Denial in Obtaining Coverage due to Health History (within past 2 years), Difficulty Finding and Choosing a Plan

Underinsurance: Not Taking a New Job in Order to Keep Health Insurance, Difficulty Finding a Provider who Accepts Insurance/ Not Able to Obtain an Appointment as Needed, Unmet Healthcare Need Due to Cost, Provider Visits in Past Year, or Out of Pocket Healthcare Costs, Out of Pocket Healthcare Costs/Premium Costs, Problems Due to Medical Expenses, Worry Related to Medical Costs

Coverage-Related Variables: Current Coverage and Coverage History

#### VII. RISKS AND DISCOMFORTS

## Psychological Risks

Individuals may find it stressful to answer questions about their experiences with health insurance coverage and care. The risks associated with these discussions are minimal, and do not rise above the level of harm encountered during daily activities.

The potential risks to subject include: 1) Discussing health insurance coverage and care and participating in a program to discuss these issues with the navigator and the patient navigator has the potential for increasing psychological vulnerability.

These risks will be described by the patient navigator and be clearly outlined in the consent form. Participants will be encouraged to discuss any concerns with the patient navigator. In the event of a psychiatric emergency, confidentiality may be suspended. If the patient navigator notes severe distress, Dr. Park will contact the participant to assess for safety and report concerns as soon as possible to the LTFU PI, Dr. Greg Armstrong, and the LTFU Project Director, Dr. Aaron McDonald, at St. Jude Children's Research Hospital. Participants will be informed of the limits of confidentiality at the beginning of the study.

#### Procedures for Minimizing Risk

Every effort will be made to minimize the study burden. The time commitment will be explained to all participants prior to the focus groups and pilot trial study consent. Every effort will be made to minimize the length and maximize the convenience or the pilot surveys completion.

#### Maintaining Confidentiality

There is a low risk that protected health information could be impermissibly disclosed or that the confidentiality of patient information may be breached. Stringent guidelines are established in order to assure the confidentiality of study subjects. A unique study identification number will serve as the primary identifier for study participants. Personal identifiers will not be part of the computerized data record. Names and addresses will be maintained in a password protected restricted data file accessible only to the principal investigator, study coordinator and designated personnel within the Data Coordinating Center. A hard copy of names and corresponding study ID numbers will be kept in a locked file cabinet within the CCSS Coordinating Center. The computerized file will only be used for generation of correspondence with the study subject. Personal identifiers will be removed from all survey booklets following completion of initial editing and scanning. Similarly, names will be removed from all LTFU abstracted information. Study participants are informed of the potential risks and benefits regarding the security of their personal information. MGH TeleHealth enables connection through virtual HIPAA-compliant videoconferencing technology including: phone, video, text, email, mobile applications and remote monitoring. These virtual visits are conducted via a Zoom videoconference platform. Zoom has been approved for use in this study by RISO review.

#### **VII. POTENTIAL BENEFITS**

The consent form for the overall LTFU study enrollment clearly states that there may be no direct benefit to the participants from study participation. For the pilot trial phase of the proposed study, participants in both groups will be given information that could improve their ability to access affordable coverage. Participants in the intervention group will also receive navigation support, for up to 4 phone-delivered sessions. As an alternative to the intervention, participants may explore health insurance support options at their current primary care center.

#### IX. MONITORING AND QUALITY ASSURANCE

Training of all Study Personnel in the Responsible Conduct of Human Studies
Prior to recruiting subjects or handling study data, all study personnel will be required to pass an NIH-approved course that reviews regulatory and informational documents on human subject protection and the responsible conduct of human studies. In addition, all study personnel will sign a statement of commitment to the protection of the rights and welfare of human subjects participating in research. In addition, all study staff must complete and submit Conflict of Interest (COI) Disclosure forms to their respective institutions.

#### Data Monitoring Plan

Survey data will be collected via Dr. Kirchhoff's team at the Huntsman Cancer Institute. Data will be collected via mailed/phone-based survey and through a secure web-based portal (REDCap). Data transmissions will be conducted between the CCSS coordinating

center and statistical center with Dr. Kirchhoff to generate the participant sample and to facilitate data access from the LTFU baseline and follow up surveys. While the majority of surveys will be done via web using REDCap, we will allow participants to complete the baseline and follow-up surveys through mail or phone to improve participation. To ensure security, participant data collected using paper and pencil records will be stored in a locked filing cabinet in a locked room at the Huntsman Cancer Institute at the University of Utah; electronic participant tracking databases will be stored on a secure server accessible only by IRB-approved members of Dr. Kirchhoff's study staff. Data collected on paper and pencil forms or through phone-based surveys will be thoroughly cleaned and entered into the electronic REDCap database with a 10% check; discrepancies will be resolved by Dr. Kirchhoff. Dr. Kirchhoff will lead the pilot study data management and analyses, and transmit analytic data to MGH using the Hartwell Center's FTA protocol (located at http://fta.stjude.org), which is a web-based interface with a secure 128-bit encrypted web connection. Only study staff will have access to the study data on Shared File Areas. Data quality (including sessions participated in for the intervention group, data missingness, and recruitment rates) will be monitored monthly. Interim data analysis will be conducted throughout the trial and results will be reported in the annual ACS progress report.

## **Adverse Events Reporting**

Serious adverse events will be reported to Drs. Park and McDonald (LTFU PI) immediately. Dr. Park will be responsible for the reporting of any adverse events to the Massachusetts General Hospital Institutional Review Board. The MGH IRB requires that serious adverse events are to be reported to the IRB as soon as possible, but no later than 10 working days from the date on which the investigator became aware of the event. Non-serious adverse events are to be reported within 20 working days. The St. Jude IRB reviews reports of unanticipated events involving risks to participants and others. The level and rapidity of review will depend upon factors such as the seriousness of the event.

#### X. REFERENCES

- 1. Robison LL, Hudson MM. Survivors of childhood and adolescent cancer: Lifelong risks and responsibilities. Nat Rev Cancer 14:61-70, 2014
- 2. Kirchhoff AC, Kuhlthau K, Pajolek H, Leisenring W, Armstrong GT, Robison, LL Park ER Employer-sponsored health insurance coverage limitations: results from the Childhood Cancer Survivor Study, 2013, Support Care Cancer
- 3. Kirchhoff AC, Nipp R, Warner EL, et al. "Job Lock" Among Long-term Survivors of Childhood CancerA Report From the Childhood Cancer Survivor Study. JAMA Oncol. Published online October 19, 2017. doi:10.1001/jamaoncol.2017.3372.
- 4. Park ER, Li FP, Liu Y, et al. Health insurance coverage in survivors of childhood cancer: The Childhood Cancer Survivor Study. J Clin Oncol 23:9187-9197, 2005

- 5. Park ER, Kirchhoff AC, Zallen JP, et al. Childhood Cancer Survivor Study participants' perceptions and knowledge of health insurance coverage: Implications for the Affordable Care Act. J Cancer Surviv 6:251-259, 2012
- 6. Oeffinger KC, Mertens AC, Hudson MM, et al. Health Care of Young Adult Survivors of Childhood Cancer: A Report from the Childhood Cancer Survivor Study. Annals of Family Medicine. 2004;2(1):61-70. doi:10.1370/afm.26.
- 7. Yeazel MW, Oeffinger KC, Gurney JG, Mertens AC, Hudson MM, Emmons KM, Chen H, Robison LL. The cancer screening practices of adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Cancer. 2004 Feb 1; 100(3): 631-640.
- 8. Casillas J, Castellino SM, Hudson MM, et al. Impact of Insurance Type on Survivor-Focused and General Preventive Health Care Utilization in Adult Survivors of Childhood Cancer: The Childhood Cancer Survivor Study (CCSS).Cancer. 2011;117(9):1966-1975. doi:10.1002/cncr.25688.
- 9. Keegan TH, Tao L, DeRouen MC, Wu XC, Prasad P, Lynch CF, Shnorhavorian M, Zebrack BJ, Chu R, Harlan LC, Smith AW, Parsons HM, AYA HOPE Study Collaborative Group. Medical care in adolescents and young adult cancer survivors: what are the biggest access-related barriers? J Cancer Surviv. 2014 Jun; 8(2): 282-292.
- 10. Kirchhoff AC, Lyles CR, Fluchel M, Wright J, Leisenring W. Limitations in health care access and utilization among long-term survivors of adolescent and young adult cancer. Cancer. 2012; 118(23): 5964-5972
- 11. Pang JW, Friedman DL, Whitton JA, et al. Employment status among adult survivors in the Childhood Cancer Survivor Study. Pediatr Blood Cancer 50:104-110, 2008
- Janson C, Leisenring W, Cox C, et al. Predictors of marriage and divorce in adult survivors of childhood cancers: A report from the Childhood Cancer Survivor Study. Cancer Epidemiol Biomarkers Prev 18:2626-2635, 2009
- 13. Kirchhoff AC, Leisenring W, Krull KR, et al. Unemployment among adult survivors of childhood cancer: A report from the Childhood Cancer Survivor Study. Med Care 48:1015-1025, 2010
- 14. Public Law 111-148, Patient Protection and Affordable Care Act. www.gpo.gov/fdsys/pkg/PLAW-111publ148/pdf/PLAW-111publ148.pdf

- 15. Mueller EL, Park ER, Davis MM. What the Affordable Care Act means for survivors of pediatric cancer. J Clin Oncol 32:615-617, 2014
- 16. Park ER, Kirchhoff AC, Perez GK, Leisenring W, Weissman JS, Donelan K, Mertens AC, Reschovsky JD, Armstrong GT, Robison LL, Franklin M, Hyland KA, Diller LR, Recklitis CJ, Kuhlthau KA. Childhood Cancer Survivor Study Participants' Perceptions and Understanding of the Affordable Care Act. Journal of Clinical Oncology.2015 March 01; 33(7): 764-772.
- 17. Warner EL, Park ER, Stroup A, Kinney AY, Kirchhoff AC. Childhood Cancer Survivors' Familiarity With and Opinions of the Patient Protection and Affordable Care Act. Journal of Oncology Practice. 2013 September 01; 9(5): 246-250
- 18. Davidoff, A. J., et al. (2015). The Affordable Care Act and Expanded Insurance Eligibility Among Nonelderly Adult Cancer Survivors. J Natl Cancer Inst. 2015;107(9).
- 19. Paez, K.A., Mallery, C.J., Noel, H., Pugliese, C., McSorely, V.E., Lucado, J.L., & Ganachari, D. (2014). Development of the Health Insurance Literacy Measure (HILM): Conceptualizing and Measuring Consumer Ability to Choose and Use Private Health Insurance. Journal of Health Communication. 2014;19(sup2): 225-239
- 20. Landier W, Bhatia S, Eshelman DA, et al: Development of risk-based guidelines for pediatric cancer survivors: The Children's Oncology Group long-term follow-up guidelines from the children's oncology group late effects committee and nursing discipline. J Clin Oncol 22:4979-4990, 2004
- 21. Long SK, Goin D. Large Racial and Ethnic Differences in Health Insurance Literacy Signal Need for Targeted Education and Outreach 2014. http://hrms.urban.org/briefs/literacy-by-race.html. Accessed Dec 2, 2014.
- 22. McCormack L, Bann C, Uhrig J, Berkman N, Rudd R. Health Insurance Literacy of Older Adults. Journal of Consumer Affairs. Summer2009 2009;43(2):223-248.
- 23. Sinaiko AD, Ross-Degnan D, Soumerai SB, Lieu T, Galbraith A. The experience of Massachusetts shows that consumers will need help in navigating insurance exchanges. Health Aff (Millwood). 2013;32(1):78-86.
- 24. Housten AJ, Furtado K, Kaphingst KA, et al. Stakeholders' perceptions of ways to support decisions about health insurance marketplace enrollment: a qualitative study. BMC Health Services Research. 2016;16:634. doi:10.1186/s12913-016-1890-8.

- 25. Pratt-Chapman M, Simon MA, Patterson A, Risendal BC, Patierno S. SURVIVORSHIP NAVIGATION OUTCOME MEASURES: A report from the ACS Patient Navigation Working Group on Survivorship Navigation. Cancer. 2011;117(15 0):3575-3584. doi:10.1002/cncr.26261.
- 26. Mulrooney DA, Yeazel MW, Kawashima T, et al. Cardiac outcomes in a cohort of adult survivors of childhood and adolescent cancer: Retrospective analysis of the childhood cancer survivor study cohort. BMJ. 2009;339:b4606.
- 27. Park ER, Kirchhoff AC, Perez GK, Leisenring W, Weissman JS, Donelan K, Hyland K, Armstrong GT, Robison LL, Kuhlthau KA. Childhood cancer survivor study participants' experiences with health insurance coverage. Society of Behavioral Medicine 36th Annual Meeting. 2015.
- 28. Kuhlthau K, Nipp RD, Shui A, et al. Health Insurance Coverage, Care Accessibility, and Affordability for Adult Survivors of Childhood Cancer: A Cross-Sectional Study of a Nationally Representative Database. Journal of Cancer Surv. 10(6): 969-971, 2016.
- 29. Park ER, Kirchhoff AC, Nipp RD, et al. Assessing Health Insurance Coverage Characteristics and Impact on Health Care Cost, Worry, and Access: A Report From the Childhood Cancer Survivor Study. JAMA Intern Med. 2017;177(12):1855–1858. doi:10.1001/jamainternmed.2017.5047
- 30. Nipp RD, Kirchoff AC, Fair D, et al. Financial Burden in Survivors of Childhood Cancer: A Report from the Childhood Cancer Survivor Study. Journal of Clinical Oncology 35(30):3474-3481, 2017.
- 31. Emmons KM, Puleo E, Park E, Gritz ER, Butterfield RM, Weeks JC, et al. Peer-delivered smoking counseling for childhood cancer survivors increases rate of cessation: the partnership for health study. J Clin Oncol 2005; 23, 6516-23.
- 32. Park ER, Puleo E, Butterfield RM, Zorn M, Mertens AC, Gritz ER, et al. A process evaluation of a telephone-based peer-delivered smoking cessation intervention for adult survivors of childhood cancer: the partnership for health study. Prev Med 2006; 42, 435-42.
- 33. Park EB, Emmons KM, Malloy NW, Seifer E. A qualitative exploration of health perceptions and behaviors among adult survivors of childhood cancers. J Cancer Educ 2002; 17, 211-5.

- 34. Butterfield RM, Park ER, Puleo E, Mertens A, Gritz ER, Li FP, et al. Multiple risk behaviors among smokers in the Childhood Cancer Survivors Study cohort. Psycho-Oncology 2004; 13, 619-629.
- 35. Duffey-Lind EC, O'holleran E, Healey M, Vettese M, Diller L, Park ER. Transitioning to survivorship: a pilot study. J Pediatr Oncol Nurs 2006; 23, 335-43.
- 36. Earle CC, Park ER, Lai B, Weeks JC, Ayanian JZ, Block S. Identifying potential indicators of the quality of end-of-life cancer care from administrative data. J Clin Oncol 2003; 21, 1133-8.
- 37. Wescott PH, Reifler EJ, Sepucha K, Park ER. Breast cancer treatment decision making: Does the sisterhood of breast cancer transcend culture? Research in the Sociology of Health Care: Health Care Services, Racial and Ethnic Minorities and Underserved Populations 2005; 23.
- 38. Bober SL, Park ER, Schmookler T, Medeiros, Nancarrow C, Diller L. Perceptions of breast cancer risk and cancer screening: a qualitative study of young, female Hodgkin's disease survivors. J Cancer Educ 2007; 22, 42-6.
- 39. Warner EL, Wu Y, Hacking CC, Wright J, Spraker-Perlman HL, Gardner E, Kirchhoff AC. Improving quality of pediatric cancer survivor care: Providers' support of and experience with survivor care plans.. Journal of Clinical Oncology. 2014; suppl 30; abstr 190.
- 40. Perrin JM, Ettner SL, Mclaughlin TJ, Gortmaker SL, Bloom SR, Kuhlthau K. State variations in supplemental security income enrollment for children and adolescents. Am J Public Health 1998; 88, 928-31.
- 41. Kuhlthau K, Perrin JM, Ettner SL, Mclaughlin TJ, Gortmaker SL. Highexpenditure children with Supplemental Security Income. Pediatrics 1998; 102, 610-5.
- 42. Perrin JM, Kuhlthau K, Ettner SL, Mclaughlin TJ, Gortmaker SL. Previous medicaid status of children newly enrolled in SSI. Health Care Financial Review 1998; 19, 117-127.
- 43. Perrin JM, Kuhlthau K, Mclaughlin TJ, Ettner SL, Gortmaker SL. Changing patterns of conditions among children receiving Supplemental Security Income disability benefits. Arch Pediatr Adolesc Med 1999; 153, 80-4.

- 44. Ettner SL, Kuhlthau K, Mclaughlin TJ, Perrin JM, Gortmaker SL. Impact of expanding SSI on Medicaid expenditures of disabled children. Health Care Financ Rev 2000; 21, 185-201.
- 45. Kuhlthau K, Ferris TG, Beal AC, Gortmaker SL, Perrin J.M. Who cares for medicaid-enrolled children with chronic conditions? Pediatrics 2001; 108, 906-12.
- 46. Cooper WO. & Kuhlthau K. Evaluating medicaid managed care programs for children. Ambul Pediatr 2001; 1, 112-6.
- 47. Perrin JM, Kuhlthau KA, Gortmaker SL, Beal AC, Ferris TG. Generalist and subspecialist care for children with chronic conditions. Ambul Pediatr 2002; 2, 462-9.
- 48. Kuhlthau K, Ferris TG, lezzoni Ll. Risk adjustment for pediatric quality indicators. Pediatrics 2004; 113, 210-6.
- 49. Kuhlthau K, Nyman RM, Ferris TG, Beal AC, Perrin JM. Correlates of use of specialty care. Pediatrics 2004; 113, e249-55.
- 50. Kuhlthau K, Ferris TG, Davis RB, Perrin JM, lezzoni LI. Pharmacy-and diagnosis-based risk adjustment for children with Medicaid. Med Care 2005; 43, 1155-9.
- 51. Kuhlthau K, Hill, KS, Fluet C, Yucel RM, Meara, E. Correlates of therapy use and expenditures in children in the United States. Developmental Neurorehabilitation,2008; 11(2):115-23.
- 52. Hill KS, Freeman LC, Yucel RM, Kuhlthau KA. Unmet Need among Children with Special Health Care Needs in Massachusetts. Matern Child Health J 2007
- 53. Tang M, Hill KS, Perrin JM, Bourdeau AA, Kuhlthau K. Medicaid managed care and the unmet need for mental health care among children with special health care needs. Health Services Research, 2008 Jun; 43(3): 882–900.
- 54. Gnanasekaran S, Arauz A, Yucel R, Hill KS, Kuhlthau K. State policy environment and delayed or forgone care among children with special health care needs. Maternal and Child Health Journal, 2008; 12(6):739-46.
- 55. Perrin JM, Fluet C, Kuhlthau KA, Anderson B, Wells N, Epstein S et al. Benefits for employees with children with ADHD: findings from the Collaborative Employee Benefit Study. J Dev Behav Pediatr 2005; 26, 3-8

- 56. Perrin JM, Fluet CF, Honberg L, Anderson B, Wells N, Epstein S et al. Benefits for employees with children with special needs: findings from the collaborative employee benefit study. Health Aff (Millwood) 2007; 26, 1096-103.
- 57. Fung V, Graetz I, Galbraith A, et al. Financial barriers to care among low-income children with asthma: Health care reform implications. JAMA Pediatrics. 2014;168(7):649-56
- 58. Galbraith AA, Ross-Degnan D, Soumerai SB, et al. Nearly half of families in high-deductible health plans whose members have chronic conditions face substantial financial burden. Health Aff (Millwood).
- 59. Galbraith AA, Soumerai SB, Ross-Degnan D, et al. Delayed and forgone care for families with chronic conditions in high-deductible health plans. J Gen Intern Med. 2012;27(9):1105-11. PMID: 22249829
- 60. Smits-Seemann RR, Kaul S, Hersh A, Fluchel M, Boucher K, Kirchhoff AC. Gaps in Insurance for pediatric patients with acute lymphoblastic leukemia. J Oncology Practice. 2016; 12(2): 175-176.
- 61. Warner EL, Kirchhoff AC, Nam G, Fluchel G. (2014). The financial burden of pediatric cancer for patients and their families. Journal of Oncology Practice. October 14.
- 62. Kirchhoff AC, Lyles CR, Fluchel M, Wright J, Leisenring W. Limitations in Health Care Access and Utilization among Adolescent and Young Adult Long-Term Cancer Survivors in the Behavioral Risk Factor Surveillance System Dataset. Cancer. 2012;118(23): 5964-72.
- 63. Galbraith AA, Sinaiko AD, Soumerai SB, Ross-Degnan D, Dutta-Linn MM, Lieu TA. Some Families Who Purchased Health Coverage Through The Massachusetts Connector Wound Up With High Financial Burdens. Health Aff (Millwood). Apr 17 2013;32(5):974-983.
- 64. Galbraith AA, Ross-Degnan D, Soumerai SB, Rosenthal MB, Gay C, Lieu TA. Nearly Half of Families In High-Deductible Health Plans Whose Members Have Chronic Conditions Face Substantial Financial Burden. Health Affairs. 2011;30(2):322-31.
- 65. Penfold RB, Kullgren JT, Miroshnik I, Galbraith AA, Hinrichsen VL, Lieu TA. Reliability of a patient survey assessing cost-related changes in health care use among high deductible health plan enrollees. BMC Health Services Research 2011, 11:133. PMCID: PMC3116474

- 66. Wisk LE, Gangnon R, Vanness DJ, Galbraith AA, Mullahy J, Witt WP.
  Development of a Novel, Objective Measure of Health Care-Related Financial
  Burden for U.S. Families with Children. Health Services Research. 2014 Oct 18
  [Epub ahead of print]
- 67. Galbraith AA, Ross-Degnan D, Soumerai S, Miroshnik I, Wharam F, Kleinman K., Lieu, TA. High-Deductible Health Plans: Are Vulnerable Families Enrolled? Pediatrics. 2009;123:e589-e594. PMCID: PMC2683628
- 68. Galbraith AA, Ross-Degnan D, Soumerai SB, Abrams AM, Kleinman K, Rosenthal MB, Wharam JF, Adams A, Miroshnik I, Lieu TA. Use of Well-Child Visits in High-Deductible Health Plans. Am J Manag Care. 2010;16(11):833-40. PMCID: PMC3984915
- 69. Lieu TA, Solomon JL, Sabin JE, Kullgren JT, Hinrichsen VL, Galbraith AA. Consumer awareness and strategies among families with high-deductible health plans. J Gen Intern Med. 2010 Mar;25(3):249-54. PMCID: PMC2839340
- 70. Wharam JF, Landon BE, Galbraith AA, Kleinman KP, Soumerai SB, Ross-Degnan D. Emergency department use and subsequent hospitalizations among members of a high-deductible health plan. JAMA. 2007:297:1093-1102.
- 71. Wharam JF, Galbraith AA, Kleinman KP, Soumerai SS, Ross-Degnan D, Landon BE. Cancer Screening among Members of a High-Deductible Health Plan. Ann Intern Med. 2008; 148: 647-655.
- 72. Balaban RB, Galbraith AA, Burns ME, Vialle-Valentin CE, Larochelle MR, Ross-Degnan D. A Patient Navigator Intervention to Reduce Hospital Readmissions among High-Risk Safety-Net Patients: A Randomized Controlled Trial. J Gen Intern Med. Jan 24 2015.
- 73. Burns ME, Galbraith AA, Ross-Degnan D, Balaban RB. Feasibility and evaluation of a pilot community health worker intervention to reduce hospital readmissions. Int J Qual Health Care. Aug 2014;26(4):358-365.
- 74. Ho W, Broughton DE, Donelan K, Gazelle GS, Hur C. Analysis of barriers to and patients' preferences for CT colonography for colorectal cancer screening in a nonadherent urban population. AJR Am J Roentgenol. 2010 Aug; 195 (2):393-7.
- 75. Donelan K, Mailhot JR, Dutwin D, Barnicle K, Oo SA, Hobrecker K, Percac-Lima S, Chabner BA. Patient perspectives of clinical care and patient navigation in follow-up of abnormal mammography. J Gen Intern Med. 2011 Feb; 26(2):116-22. Epub 2010 Jul 7.

- 76. Donelan K, Rao SR, Rogers RS, Mailhot JR, Galvin R. Experience with health coach-mediated physician referral in an employed insured population. J Gen Intern Med. 2010 Oct; 25(10):1071-7. Epub 2010 Jun 16.
- 77. Zuckerman KE, Cai X, Perrin JM, Donelan K. Incomplete specialty referral among children in community health centers. J Pediatr. 2011 Jan; 158(1):142-8.
- 78. Leon AC, Davis LL, Kraemer HC. The Role and Interpretation of Pilot Studies in Clinical Research. J Psychiatr Res. 2011 May; 45(5): 626–629.
- 79. Freund KM, Battaglia TA, Calhoun E, Dudley DJ, Fiscella K, Paskett E, Raich PC, Roetzheim RG, Patient Navigation Research Program Group. National Cancer Institute Patient Navigation Research Program: methods, protocol, and measures. Cancer. 2008 Dec 15; 113(12): 3391-3399.
- 80. Calhoun EA, Whitley EM, Esparza A, Ness E, Greene A, Garcia R, Valverde PA. A National Patient Navigator Training Program. Health Promotion Practice. 2010 March 01; 11(2): 205-215.
- 81. Oeffinger KC, Mertens AC, Sklar CA, et al. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med 355:1572-1582, 2006
- 82. Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. 1991; 32(6): 705-714.
- 83. Kornblith AB, Dowell JM, Herndon JE,2nd, Engelman BJ, Bauer-Wu S, Small EJ, Morrison VA, Atkins J, Cohen HJ, Holland JC. Telephone monitoring of distress in patients aged 65 years or older with advanced stage cancer: a cancer and leukemia group B study. Cancer. 2006 Dec 1; 107(11): 2706-2714.
- 84. Naughton MJ, Herndon JE,2nd, Shumaker SA, Miller AA, Kornblith AB, Chao D, Holland J. The health-related quality of life and survival of small-cell lung cancer patients: results of a companion study to CALGB 9033. Qual Life Res. 2002 May; 11(3): 235-248.
- 85. Queenan JA, Feldman-Stewart D, Brundage M, Groome PA. Social support and quality of life of prostate cancer patients after radiotherapy treatment. Eur J Cancer Care (Engl). 2009 Jun 22.
- 86. Bagley N, Jones DK, Jost TS. Predicting the Fallout from King v. Burwell Exchanges and the ACA. NEJM 2015;372(2):101-104
- 87. Johnson R.B., Onwuegbuzie, A. J. Mixed methods research: a paradigm whose time has come. Educational Researcher 2004; 33, 14-26.

- 88. CDC/National Center for Health Statistics: National Health Interview Survey (NHIS). http://www.cdc.gov/nchs/nhis.htm
- 89. Child and Adolescent Health Measurement Initiative: National Survey of Children with Special Health Care Needs, 2012. http://www.childhealthdata.org/learn/NS-CSHCN
- 90. Agency for Healthcare Research and Quality, US Department of Health and Human Services: Medical expenditure panel survey (MEPS), 2009. http://meps.ahrq.gov/mepsweb/
- 91. Center for Studying Health System Change (HSC): Community tracking study (CTS) and health tracking surveys. http://www.hschange.org/index.cgi?data=12
- 92. The Commonwealth Fund: Kaiser/Commonwealth 1997 National Survey of Health Insurance, 1997. http://www.commonwealthfund.org/publications/surveys/1996/kaiser-commonwealth-1997-national-survey-of-health-insurance